CLINICAL TRIAL: NCT04218760
Title: Pain Perception, Headache Provocation and Multiomics of People Who Are Unable to Have Headache
Brief Title: Multiomics After Headache Provocation of People Who Are Unable to Have Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Isa Amalie Olofsson, Principal Investigator, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HR003 Multiomics Provocation
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Headache; Healthy
MeSH Terms: conditions — Headache | interventions — isosorbide-5-mononitrate; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Case-control study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isosorbide mononitrate (Experimental): Cases and controls both receive one tablet Imdur® 60 mg (isosorbide mononitrate) on the study day and have 3 sets of blood samples drown.
  Interventions: Drug: Isosorbide Mononitrate 60 MG Extended Release Oral Tablet [Imdur]; Other: Blood sample

INTERVENTIONS:
Drug: Isosorbide Mononitrate 60 MG Extended Release Oral Tablet [Imdur] — 1 tablet Isosorbide Mononitrate 60 mg administrated orally.
Other: Blood sample — 3 blood samples from a periferal vein, two for RNA and one for metabolomics are taken right before administration of isosorbide mononitrate, 3 hours after administration of isosorbide mononitrate and again 5 hours after administration of isosorbide mononitrate.

SUMMARY:
Headaches are extremely common illnesses with a combined lifetime prevalence of 90-99% in Europe. Despite this high prevalence, there are persons who have never, in their whole life, encountered a headache.

The aim of the study is to identify factors that protect against headache by studying multiomics in people who never have had a headache (headache resistant) versus non-resistant controls.

The investigators will measure multiomic changes (transcriptomics and metabolomics) after headache provocation with isosorbide mononitrate. 3 blood samples, two for RNA and one for metabolomics are taken right before administration of isosorbide mononitrate, 3 hours after administration of isosorbide mononitrate and again 5 hours after administration of isosorbide mononitrate.

The investigators hope to contribute with novelty to the current understanding of headache pathophysiology and development of more efficient treatment of headache.

ELIGIBILITY:
Inclusion Criteria:

* Headache resistant and non-resistant male participants from the Danish Blood Donor Study.
* Weight: 45 kg to 95 kg

Exclusion Criteria:

* Daily consumption of any medication.
* Consumption of any medication less than 12 hours prior to the study day.
* Headache on the study day or 48 hours prior to the study day.
* Amnestic or clinical signs of hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) or hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg).
* Any severe cardiovascular disease, including cerebrovascular illness.
* Amnestic or clinical signs of current mental illness.
* Amnestic or clinical signs of current substance or drug abuse.
* Amnestic or clinical signs of any illness the responsible doctor considers relevant for participation in the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Transcriptomic changes | 5 hours
  Difference in RNA expression between cases and controls after headache provocation by Isosorbide Mononitrate.
Metabolomic changes | 5 hours
  Difference in metabolites between cases and controls after headache provocation by Isosorbide Mononitrate.

CONTACTS AND LOCATIONS:
Overall Officials: Jes Olesen, Professor, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Region H, Denmark

IPD SHARING:
Plan to Share IPD: Undecided